CLINICAL TRIAL: NCT07104097
Title: Regional Anesthesia in Hip Arthroplasty- Comparison Between Two Techniques for Erector Spinae Plane Block
Brief Title: Comparison Between 2 Techniques for Lumbar-ESPB
Acronym: ESPTA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Dario Bugada, MD, Papa Giovanni XXIII Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0018028/25
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hip Surgery
Keywords: erector spinae plane block; hip surgery; sensory block; motor block; local anesthetic
MeSH Terms: interventions — Anesthesia, Spinal; Dexamethasone; Ibuprofen; Acetaminophen; Morphine

STUDY DESIGN:
Intervention Model Description: randomized trial, single blind
Who Masked: Outcomes Assessor
Masking Description: outcome assessor will not be aware of the technique used in the OR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- superficial ESPB (Active Comparator): Injection on top of L3 transverse process, plane between bone and erector spinae muscle
  Interventions: Procedure: spinal anesthesia; Procedure: superficial erector spinal plane block (ESPB); Drug: Dexamethasone; Drug: Ibuprofen 400 mg; Drug: Paracetamol; Drug: Morphine
- deep ESPB (Experimental): Injection BETWEEN L3 and L4 transverse process, fascial plane between erector spinae muscle AND the deep muscles
  Interventions: Procedure: spinal anesthesia; Procedure: deep (inter laminar) erector spinal plane block (ESPB); Drug: Dexamethasone; Drug: Ibuprofen 400 mg; Drug: Paracetamol; Drug: Morphine

INTERVENTIONS:
Procedure: spinal anesthesia — spinal anesthesia at L3-L4 plain bupivacaine 0.5% 2.2 ml
Procedure: superficial erector spinal plane block (ESPB) — Lidocaine 1% + ropivacaine 0.25% 30 ml with adrenaline 1:200.000 on top of L3 transverse process, between bone and erector spinae muscle
  Arms: superficial ESPB
Procedure: deep (inter laminar) erector spinal plane block (ESPB) — Lidocaine 1% + ropivacaine 0.25% 30 ml with adrenaline 1:200.000 between L3 and L4 transverse process, between erector spinae muscle and deep muscles
  Arms: deep ESPB
Drug: Dexamethasone — 8 mg iv preoperatively
Drug: Ibuprofen 400 mg — preoperatively and postoperatively (every 8 hours)
Drug: Paracetamol — 1000 mg preoperatively and postoperatively (every 8 hours)
Drug: Morphine — Patient Controlled Analgesia

SUMMARY:
Diffusion of local anesthetics after a lumbar ESPB within fascial planes towards nerve structures is a matter of debate.

The main objective of the study is to compare the incidence of sensory block between two techniques of needle placement (superficial or translaminar) during lumbar ESPB block.

Patients are treated with lumbar ESPB (randomized to superficial or translaminar), spinal anesthesia and multimodal analgesia.

The primary endpoint will be the incidence of numbness/reduced skin sensitivity to cold (ice test) in the area innervated by the lumbar plexus. Secondary outcomes are pain and analgesic's consumption, motor block, quality of recovery and discharge ability.

ELIGIBILITY:
Inclusion Criteria:

* primary total hip replacement
* informed consent

Exclusion Criteria:

* allergies to study drugs
* spinal anesthesia contraindicated
* kidney failure (GFR<30)
* epilepsy, psychiatric disease, neurologic deficits
* revision surgery
* neuropathies in the lumbar area (tingling, hypoestesia, numbness, motor deficit)
* no informed consent
* pregnancy
* alcohol/opioid abuse
* emergency surgery/intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
sensory block | 24 hours
  incidence of reduced or abolished cold sensation on the skin in the territory of lumbar plexus (anterior, medial and lateral thigh)

SECONDARY OUTCOMES:
motor block | 24 hours
  block of extension and/or adduction of the thigh
postoperative pain | 48 hours
  numeric rating scale - NRS 11 point scale from 0 = "no pain" to 10 = "worst imaginable pain"
morphine consumption | 24 hours
  milligrams of morphine by patient controlled analgesia intravenously
quality of recovery | 48 hours
  QoR-15 (Quality of Recovery 15 items) questionnaire - global measure of postoperative recovery, with a score ranging from 0 (extremely poor) to 150 (excellent)
complications | 48 hours
  presence of nausea and vomiting, any other complication
discharge ability | 48 hours
  PADDs score (Post Anaesthetic Discharge Scoring System) - 5 items, each scored from 0 to 2, where the higher the score (from 0 to 10), the greater the degree of the patient's recovery and readiness to be discharged. Scores of 9 or 10 mean the patient can be safely discharged.

CONTACTS AND LOCATIONS:
Locations (1):
- Aast Papa Giovanni Xxiii, Bergamo, Italy